CLINICAL TRIAL: NCT03567876
Title: Rituximab, Bendamustine and Cytarabine Followed by Venetoclax (V-RBAC) in High-risk Elderly Patients With Mantle Cell Lymphoma (MCL)
Brief Title: Rituximab, Bendamustine and Cytarabine Followed by Venetoclax in High Risk Elderly Patients With MCL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIL_V-RBAC
Record Dates: First submitted 2018-05-22; First posted 2018-06-26 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Lymphoma, Mantle-Cell
Keywords: Mantle cell lymphoma; Elderly patients; First line
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- V-RBAC (RBAC followed by Venetoclax) (Experimental): Induction phase: RBAC --> up to 6 cycles for low risk (LR) patients and up to 4 cycles for high risk (HR) patients.
  Patients proceeding to Venetoclax treatment will receive consolidation with single agent Venetoclax 800 mg/die x 4 28d cycles (with initial ramp-up dose) of each consolidation cycle. Consolidation will be followed by maintenance with single agent Venetoclax 400 mg/die (V maint ) for a total of 2 years (4 months consolidation+20 months maintenance).
  Interventions: Drug: Venetoclax

INTERVENTIONS:
Drug: Venetoclax — Consolidation and maintenance phases with Venetoclax (for a total of 2 years) after an induction phase R-BAC (up to 6 cycles for law risk patients and up to 4 cycles for high risk patients)
  Other Names: Venclyxto (commercial name)

SUMMARY:
Prospective, multicenter, phase II trial designed to evaluate whether the addition of Venetoclax after rituximab, bendamustine and cytarabine (R-BAC) to high risk patients with mantle cell lymphoma improves the results of the standard R-BAC, in terms of Progression Free Survival.

DETAILED DESCRIPTION:
The aim of the study is to improve long term results of R-BAC, consolidating patients with high-risk (HR) features (defined as: elevated Ki67 and/or blastoid cytology and/or TP53 mutation after central pathology review) with Venetoclax (ABT-199), which has demonstrated relevant single agent activity in relapsed/refractory MCL in a Phase 1-2 trial.

The updated Progression Free Survival curves of the R-BAC500 trial has shown that the expected 2-years PFS for patients with HR disease is 40% (H0), as compared to low-risk patients (LR) that have a 2-years PFS of 100%. The addition of Venetoclax to HR patients after R-BAC is expected to improve results and efficacy of this regimen in this "difficult -to- treat" population, that represents approximately 40-45 % of newly diagnosed elderly patients with MCL. It appears reasonable to treat with the experimental drug also LR patients that do not respond appropriately (less than CR) at the end of R-BAC. Since the number of such LR patients is hardly predictable based on the present experience with R-BAC500 trial, the analysis of this sub-cohort will be of exploratory nature, and thus assessed separately.

The study objective is to evaluate whether the addition of venetoclax after R-BAC to HR patients improves the results of the standard R-BAC, in terms of Progression Free Survival .

ELIGIBILITY:
Inclusion Criteria:

1. Previously untreated patients with MCL aged ≥65 years if they are FIT according to the geriatric CGA assessment.
2. age ≤64 years not eliglible to high-dose chemotherapy plus transplantation at physician's judgement (details for non eligibility to be recorded by means of the CIRS, Cumulative Illness rating Scale).
3. Measurable nodal or extranodal disease ≥ 1.5 cm in longest diameter, and measurable in 2 perpendicular dimensions.
4. ECOG performance status ≤2.
5. Positivity for cyclin D1 and/or SOX11 [the latter being mandatory in cases lacking cyclin D1- or t(11;14)-negative].
6. Adequate renal function (Creatinine clearance >50 mL/min), with preserved diuresis.
7. Adequate liver function: alanine aminotransferase (ALT)/aspartate aminotransferase (AST) <2.5 x upper limit of normal (ULN) value, total bilirubin <1.5 x ULN, unless directly attributable to the patient's tumor or to congenital causes.
8. Hepatitis B core antibody (HBcAb) positive/HBsAg negative/HBV-DNA negative patients may be enrolled if correct antiviral prophylaxis is administered at least 2 weeks before initiating protocol treatment.
9. Written informed consent.

Exclusion Criteria:

1. Human immunodeficiency virus (HIV) positive.
2. Previous treatment for lymphoma.
3. Disease confined to the bone marrow/peripheral blood/spleen, without any other nodal or extranodal involvement.
4. In-situ MCL.
5. Medical conditions or organ injuries that could interfere with administration of therapy.
6. Active bacterial, viral, or fungal infection requiring systemic therapy.
7. Seizure disorders requiring anticonvulsant therapy.
8. Severe chronic obstructive pulmonary disease with hypoxiemia.
9. History of severe cardiac disease: New York Heart Association (NYHA) functional class III-IV, myocardial infarction within 6 months, ventricular tachyarrhythmias, dilatative cardiomyopathy, or unstable angina.
10. Uncontrolled diabetes mellitus.
11. Active secondary malignancy.
12. Known hypersensitivity or anaphylactic reactions to murine antibodies and proteins, to Bendamustine or mannitol.
13. Major surgery within 4 weeks of study Day 1.
14. HBsAg+
15. HCVAb+ patients with active viral replication (HCV-RNA+ with AST>2 x normal limit)
16. Any co-existing medical or psychological condition that would preclude participation in the study or compromise the patient's ability to give informed consent, or that may affect the interpretation of the results, or render the patient at high risk from treatment complications.
17. CNS involvement
18. Chronic treatment with strong or moderate CYP3A inhibitors (e.g. ketoconazole, ritonavir, clarithromycin, itraconazole, voriconazole)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2021-07-26 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Progression-free survival of the High Risk patients | 24 months
  2-years progression-free survival (PFS) of the HR patients from date of enrollment

SECONDARY OUTCOMES:
Molecular response | 10 months and 30 months
  The proportion of molecular response (analyzed in the labs of the FIL- MRD Network)
Progression-free survival of all patients and different subgroups | 24 months
  The progression-free survival (PFS) of all enrolled patients, and of different subgroups (i.e TP53 mutated patients)
Overall survival | 54 months
  Overall survival
Duration of responses | 24 months
  Duration of responses
Proportion of complete remission in High Risk and Law Risk patients | 6 months and 10 months
  The proportion of complete remission (CR) before and after venetoclax in the HR group and/or in the LR not responding to R-BAC
Completed expected treatment schedule | 30 months
  The proportion of patients that complete the expected treatment schedule
Incidence of Treatment-Emergent Adverse Events | 10 months and 30 months
  The proportion of patients with adverse events as assessed by CTCAE 4.03 during venetoclax administration as consolidation or maintenance after R-BAC

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Visco, MD, Principal Investigator — AOU Integrata di Verona - U.O. Ematologia -Verona -Italy
Locations (35):
- Italy (35):
  - A.O. SS. Antonio e Biagio e Cesare Arrigo, SC Ematologia, Alessandria
  - Università Politecnica delle Marche, Clinica di Ematologia, Ancona
  - Centro Riferimento Oncologico, S.O.C. Oncologia Medica A, Aviano
  - IRCCS Istituto Tumori Giovanni Paolo II, UOC Ematologia, Bari
  - Policlinico S. Orsola-Malpighi, Istituto di Ematologia "Seragnoli", Bologna
  - ASST Spedali Civili, Ematologia, Brescia
  - Ospedale Businco, Ematologia, Cagliari
  - Azienda Ospedaliera S. Croce e Carle, SC Ematologia, Cuneo
  - Azienda Ospedaliera Universitaria Careggi, Unità funzionale di Ematologia, Florence
  - Ospedale Policlinico San Martino S.S.R.L. - IRCCS per l'Oncologia, Clinica Ematologica, Genova
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (I.R.S.T.), Ematologia, Meldola
  - ASST Grande Ospedale Metropolitano Niguarda, SC Ematologia, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori di Milano, Ematologia, Milan
  - Istituto Scientifico San Raffaele, Unità Linfomi - Dipartimento Oncoematologia, Milan
  - Ospedale Maggiore Policlinico - Fondazione IRCCS Ca' Granda, Ematologia, Milan
  - AOU Maggiore della Carità di Novara, SCDU Ematologia, Novara
  - Azienda Ospedaliera Universitaria di Padova, Ematologia, Padua
  - A.O. Ospedali Riuniti Villa Sofia-Cervello, Divisione di Ematologia, Palermo
  - IRCCS Policlinico S. Matteo, Divisione di Ematologia, Pavia
  - Ospedale Guglielmo Da Saliceto, UO Ematologia, Piacenza
  - Ospedale delle Croci, Ematologia, Ravenna
  - Grande Ospedale Metropolitano Bianchi Melacrino Morelli, Ematologia, Reggio Calabria
  - Azienda Unità Sanitaria Locale-IRCCS - Arcispedale Santa Maria Nuova, Ematologia, Reggio Emilia
  - Ospedale degli Infermi, UO Ematologia, Rimini
  - Policlinico Umberto I - Università "La Sapienza", Istituto Ematologia -Dipartimento di Biotecnologie Cellulari ed Ematologia, Roma
  - Università Cattolica S. Cuore, Ematologia, Roma
  - Istituto Clinico Humanitas, UO Ematologia, Rozzano
  - A.O.U. Città della Salute e della Scienza di Torino, SC Ematologia Universitaria, Torino
  - A.O.U. Città della Salute e della Scienza di Torino, SC Ematologia, Torino
  - Ospedale Ca' Foncello, SC Ematologia, Treviso
  - Azienda Ospedaliera C. Panico, UOC Ematologia e Trapianto, Tricase
  - Azienda Sanitaria Universitaria Integrata di Udine, Clinica Ematologica, Udine
  - Ospedale di Circolo, UOC Ematologia, Varese
  - Azienda Ospedaliera Universitaria Integrata di Verona, UO Ematologia, Verona
  - Ospedale San Bortolo, Divisione di Ematologia, Vicenza

REFERENCES:
- [Derived] Visco C, Tabanelli V, Sacchi MV, Evangelista A, Quaglia FM, Fiori S, Bomben R, Tisi MC, Riva M, Merli A, Rotondo F, Fraenza C, Carazzolo ME, Corradini P, Farina L, Castellino C, Castellino A, Zilioli VR, Muzi C, Piazza F, Re A, Hohaus S, Rossi FG, Musuraca G, Di Rocco A, Puccini B, Sciarra R, Ballerini F, Cavallo F, Bruna R, Moia R, Moioli A, Bernardelli A, Drandi D, Arcari A, Merli F, Gini G, Freilone R, Tani M, Pavone V, Ladetto M, Pileri SA, Balzarotti M; Fondazione Italiana Linfomi. Rituximab, bendamustine, and cytarabine followed by venetoclax in older patients with high-risk mantle cell lymphoma (FIL_V-RBAC): a multicentre, single-arm, phase 2 study. Lancet Haematol. 2025 Oct;12(10):e777-e788. doi: 10.1016/S2352-3026(25)00252-2. Epub 2025 Sep 17. PMID 40975105